CLINICAL TRIAL: NCT03052361
Title: Triage Administration of Ondansetron for Gastroenteritis in Children; a Randomized Controlled Trial
Brief Title: Triage Administration of Ondansetron for Gastroenteritis in Children
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The recruitment was much slower than expected and the COVID pandemic added new barriers to recruitment.
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, Principal investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ondansetron at triage
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Gastroenteritis
Keywords: Children; emergency department; ondansetron
MeSH Terms: conditions — Gastroenteritis; Emergencies | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron (Experimental): Patients allocated to this arm will receive ondansetron in the ED triage. Posology of ondansetron will be adapted to weight: doses of 2 mg for children weighting between 8 and 15 kg, 4 mg for children weighting between 15 to 30 kg and 8 mg for children heavier than 30 kg
  Interventions: Drug: Ondansetron
- control (Placebo Comparator): Patients allocated to this arm will receive an identical looking/tasting placebo in the ED triage.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ondansetron — Patients allocated to this arm will receive ondansetron in the ED triage.
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebos — similar looking and tasting liquid placebo
  Arms: control

SUMMARY:
The investigators aim to assess whether ondansetron given at triage can reduce the number of patients requiring emergency department observation in children with acute gastroenteritis. The investigators will also assess the improvement of patient comfort and total length of stay

DETAILED DESCRIPTION:
Background:

Acute gastroenteritis is one the most common cause of emergency room visits. Studies have demonstrated that ondansetron is effective in reducing vomiting in children with gastroenteritis and improve outcomes by decreasing intravenous rehydration and hospital admission of those patients. Giving ondansetron to children with suspected gastroenteritis immediately at triage could reduce the number of patients requiring observation in the emergency department after medical consultation and improve patients' outcomes.

Objective:

The aim of this study is to assess the effectiveness of triage-initiated administration of ondansetron for suspected gastroenteritis in the paediatric emergency department. The investigators aim to assess whether ondansetron given at triage can reduce the number of patients requiring observation in children with acute gastroenteritis. The investigators will also assess the improvement of patient comfort and total length of stay.

Methods:

This will be a randomized controlled trial performed in a tertiary paediatric emergency department. Participants will include all infants more than 8kg who present to the emergency department with at least four vomiting in the previous 24 hours and the last vomiting that occurred in the previous 2h. The intervention will consist of giving ondansetron at triage versus placebo. The primary outcome will be the number of patients requiring observation after medical consultation in both groups. Secondary objectives will be the number of episodes of vomiting after receiving the intervention, length of stay in the emergency department and the proportion of children who will return to a physician within 48 hours. The investigators will assess the improvement of patient comfort evaluated by parents according to a BARF (Baxter Animated Retching Face) Scale within the ondansetron group vs placebo. The primary analysis will be the comparison of the proportion of observation for the two groups. Based on a preliminary study of the currents children suffering from gastro-enteritis, it was estimated that the recruitment of 248 participants will provide a power of 90% to identify a 20% difference in the proportion of observed patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged more than 6 months and weight ≥ 8kg
* At least 4 non-bilious, non-bloody vomiting in the preceding 24 hours
* The last vomiting occured less than 2 hours ago
* No other diagnostic more likely than gastroenteritis suspected by the nurse at triage.

Exclusion Criteria:

* Severe dehydration (based on poor capillary refill or hypotension)
* Underlying disease that could affect the assessment of hydration (such as renal failure or hypoalbuminemia)
* Bilious or bloody vomiting
* Bloody stool
* A history of abdominal surgery
* Allergy to ondansetron
* Long QT syndrome or major cardiac condition
* Previous enrolment in the study.
* Girl at risk of pregnancy (pubertal girl)
* Inability to obtain parental informed consent (language barrier, absence, etc.)

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-10-03 (Actual)

PRIMARY OUTCOMES:
Disposition | 12 hours
  The number of patients that are discharged immediately after initial medical assessment

SECONDARY OUTCOMES:
Length of Stay | 12 hours
  The ED length of stay from registration to discharged
ED vomiting | 12 hours
  The number of episodes of vomiting in the ED.
48 hours vomiting | 48 hours
  The number of episodes of vomiting in the 24 and 48 hours
Return visit | 48 hours
  The number of patients who return to ED and to a physician within 48 hours.
Nausea level | 12 hours
  Improvement of patient comfort evaluated by parents according to a Baxter Animated Retching Face Scale (BARF) scale
Alternative diagnosis | 12 hours
  In a safety analysis, the investigator will evaluate if the nurse at triage was correct in suspecting that the enrolled children were suffering from gastroenteritis and we will compare the proportion of alternate diagnosis in both groups
Left without being sen | 12 hours
  The investigator will compare the proportion of children who left the ED without being seen by a physician.
Rescue medication | 12 hours
  The proportion of children requiring a rescue medication for persistent nausea/vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, Principal Investigator — Sainte-Justine Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No